CLINICAL TRIAL: NCT01045811
Title: Effects of Breathing Training on Psychosocial Functioning and Heart Rate Variability in Postmenopausal Women With Depressive Symptoms-3
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were recruited at this study site. Study has been conducted and monitored with ClinicalTrials.gov ID: NCT01044563.
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pei-Shan Tsai, Professor, College of Nursing, Taipei Medical University, National Science and Technology Council, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC98-2629-B-038-002-MY3-WFH
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Postmenopause
Keywords: Depression; Depressive Symptoms; postmenopause; RSA biofeedback
MeSH Terms: conditions — Depression | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breathing training (Experimental): Respiratory sinus arrhythmia biofeedback-assisted deep breathing training
  Interventions: Behavioral: Breathing training
- Stress management (Active Comparator): Cognitive reconstructive strategies for stress management
  Interventions: Behavioral: Stress management

INTERVENTIONS:
Behavioral: Breathing training — Respiratory sinus arrhythmia biofeedback-assisted deep breathing training
  Arms: Breathing training
Behavioral: Stress management — Cognitive reconstructive strategies for stress management
  Arms: Stress management

SUMMARY:
The specific aims of this study are:

1. To develop a breathing training protocol specifically designed to improve HRV and psychosocial functioning for postmenopausal women with depressive symptoms,
2. To examine the immediate effects of an 8-week breathing training program on HRV and psychosocial end points in postmenopausal women with depressive symptoms,
3. To examine the intermediate-term effects of an 8-week breathing training program on HRV and psychosocial end points in postmenopausal women with depressive symptoms, and
4. To determine whether the change in depressive symptoms with breathing training in postmenopausal women is associated with the change in HRV.

DETAILED DESCRIPTION:
Postmenopausal women without hormone replacement therapy are associated with higher risk of cardiac morbidity and mortality. They are likely to experience depressive symptoms after menopause, and the comorbidity of depression are related to altered autonomic function. We expect that postmenopausal women with depressive symptoms who receive breathing training will demonstrate decreased depressive symptoms and increased heart rate variability immediately upon and later after completion of training, and optimally contributing to improve autonomic nervous regulation in their later life to prevent undesired cardiac outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Permanent termination of menstruation of natural cause.
* Cessation of menstrual cycles for more than 12 consecutive months.
* A score of the Chinese version of Beck Depression Inventory-II of greater than 10.
* Able to speak Mandarin or Taiwanese.
* Age from 45 to 64 years.

Exclusion Criteria:

* Subjects who are clinically diagnosed with history of cardiac arrhythmia, coronary heart disease, heart failure, kidney disease, hypertension, chronic low blood pressure, diabetic neuropathy, psychosis, mental deficiency.
* Subjects who received hormone replacement therapy prescribed by gynecological physicians.
* Subjects who took cardiac and/or psychotropic medications which may affect the autonomic functions

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05

PRIMARY OUTCOMES:
Depressive symptoms | baseline
Depressive symptoms | posttest (8 weeks from baseline)
Depressive symptoms | follow-up (16 weeks from baseline)

SECONDARY OUTCOMES:
Heart rate variability (Resting, reactivity to stress, and recovery from stress) | baseline
Heart rate variability (Resting, reactivity to stress, and recovery from stress) | posttest (8 weeks from baseline)
Heart rate variability (Resting, reactivity to stress, and recovery from stress) | follow-up (16 weeks from baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Wangfang Hospital, Taipei, Wenshan Dist., Taiwan